CLINICAL TRIAL: NCT02591290
Title: Immunogenicity and Safety of Two-Dose Series of a Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (SP284; Menactra®) in Japanese Healthy Adult Subjects
Brief Title: Immunogenicity and Safety of Two-Dose Series of Menactra® in Japanese Healthy Adult Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EFC14375/MTA89; U1111-1174-4291 (Other: WHO)
Record Dates: First submitted 2015-10-27; First posted 2015-10-29 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Meningitis; Meningococcal Meningitis; Meningococcal Infections
Keywords: Meningitis; Meningococcal Meningitis; Meningococcal Infections; Menactra®; Meningococcal Vaccine
MeSH Terms: conditions — Meningitis; Meningitis, Meningococcal; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Menactra® Vaccine (Experimental): Participants received 2-dose series of the study vaccine with 8-week interval.
  Interventions: Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate

INTERVENTIONS:
Biological: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular (2 doses with 8-week interval)
  Other Names: SP284; Menactra®

SUMMARY:
The aim of this study was to collect further information regarding an increase immune response of SP284 after an additional dose in Japanese participants.

Primary Objective:

* To evaluate and describe the immune responses to meningococcal antigens (serogroups A,C, Y and W-135) at 28 days following each vaccination with SP284 vaccine in participants 20 through 55 years of age.

Other Pre-specified objective:

* To describe the safety in terms of immediate systemic adverse events (AEs), solicited reactions, unsolicited non-serious adverse events, and serious adverse events (SAEs) following receipt of each dose of SP284 vaccine in persons 20 through 55 years of age.

DETAILED DESCRIPTION:
All participants received a 2-dose series of the study vaccine with 8-week interval and was monitored for safety and assessed for immunogenicity at baseline (pre-vaccination) and at 28 to 35 days following each vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 through 55 years on the day of inclusion,
* Informed consent form had been signed and dated by the participant,
* Able to attend all scheduled visits and to comply with all trial procedures,
* For female participants who had childbearing potential, use of an effective method of contraception from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination
* a) "20 through 55 years" meant from the day of the 20th birthday to the day before the 56th birthday.
* b) To be considered to be not of childbearing potential, a woman must either had undergone surgical sterilization (hysterectomy or bilateral tubal ligation) or be postmenopausal (at least one year without menses) at the time of vaccination. Effective methods of contraception include oral contraception (pill), intrauterine device, diaphragm or condoms used with sponge, contraceptive foam or cream, hormonal implants, transdermal patch, or parenteral contraception.

Exclusion Criteria:

* Chronic illness that, in the opinion of the investigator, was at a stage where it might interfere with trial conduct or completion,
* History of meningococcal diseases, confirmed either clinically, serologically, or microbiologically,
* Known systemic hypersensitivity to any of the vaccine components, or history of a life threatening reaction to a vaccine containing the same substances of the study vaccine,
* Known or suspected congenital or current/ previous acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroids therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months),
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the trial inclusion,
* Planned participation in another clinical trial during the present trial period,
* Receipt of immune globulins, blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response,
* Receipt of any vaccine within the four weeks preceding the trial vaccination, except for influenza vaccination, which might be received at least two weeks before the study vaccine,
* Planned receipt of any vaccine during the trial period,
* Clinical or known serological evidence of systemic illness including Hepatitis B, Hepatitis C and/or Human Immunodeficiency Virus infection,
* Participant was pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination and until at least 4 weeks after the last vaccination),
* Known thrombocytopenia, contraindicating intramuscular (IM) vaccination,
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination,
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily,
* Current alcohol abuse or drug addiction,
* Identified as employee of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family member (i.e., immediate, husband, wife and their children, adopted or natural) of the employees or the Investigator,
* Previous vaccination against meningococcal disease with either the trial vaccine or another vaccine,
* At high risk for meningococcal infection during the trial,
* Febrile illness (temperature ≥ 37.5°C) or moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination. A prospective participant should not be included in the study until the condition had resolved or the febrile event had subsided,
* Received oral or injected antibiotic therapy within the 72 hours prior to blood draw (Visit 1),
* History of Guillain-Barré Syndrome (GBS).

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2016-03-16 (Actual); Study Completion 2016-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi KK
Locations (1):
- Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 20 October 2015 through 18 December 2015 at a single center in Japan.
Pre-assignment Details: A total of 60 participants were enrolled in the study.
Groups:
- Menactra® Vaccine: Participants received 2 doses of 0.5 mL Menactra® Vaccine, intramuscularly, with 8-week interval.
Period: Overall Study
Arm/Group | Menactra® Vaccine
Started | 60
Vaccinated Dose 1 | 60
Vaccinated Dose 2 | 58
Completed | 58
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Menactra® Vaccine
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 32
Region of Enrollment [Number; unit: participants]
  Japan | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Meningococcal Serogroups A, C, Y, and W-135 Antibody Titers >=1:128
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by Serum Bactericidal Assay using Baby Rabbit complement (SBA-BR).
Time Frame: Day 0 (pre-vaccination), Day 28 post-vaccination 1, Day 28 post-vaccination 2
Population: Per Protocol (PP) analysis set included all participants who received 2 study vaccinations and provided the valid blood samples of pre-vaccination and post-1st and post-2nd vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Menactra® Vaccine
Number analyzed (Participants) | 56
Participants
  Serogroup A (Pre-Vaccination) | 43
  Serogroup A (Day 28 post-vaccination 1) | 56
  Serogroup A (Day 28 post-vaccination 2) | 56
  Serogroup C (Pre-Vaccination) | 15
  Serogroup C (Day 28 post-vaccination 1) | 47
  Serogroup C (Day 28 post-vaccination 2) | 52
  Serogroup Y (Pre-Vaccination) | 28
  Serogroup Y (Day 28 post-vaccination 1) | 54
  Serogroup Y (Day 28 post-vaccination 2) | 53
  Serogroup W-135 (Pre-Vaccination) | 15
  Serogroup W-135 (Day 28 post-vaccination 1) | 51
  Serogroup W-135 (Day 28 post-vaccination 2) | 53

2. Other Pre Specified Outcome: Number of Participants With >=4-Fold Rise in Meningococcal Serogroups A, C, Y, and W-135 Antibody Titers Following Vaccination
Description: Meningococcal serogroups A, C, Y, and W-135 antibody titers were measured by SBA-BR in the serum specimens. Number of participants with >=4-fold rise in each meningococcal serogroups antibody titer at Day 28 post-vaccination 1 and at Day 28 post-vaccination 2 were reported.
Time Frame: Day 28 post-vaccination 1, Day 28 post-vaccination 2
Population: PP analysis set included all participants who received 2 study vaccinations and provided the valid blood samples of pre-vaccination and post-1st and post-2nd vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Menactra® Vaccine
Number analyzed (Participants) | 56
Participants
  Serogroup A (Day 28 post-vaccination 1) | 40
  Serogroup A (Day 28 post-vaccination 2) | 39
  Serogroup C (Day 28 post-vaccination 1) | 46
  Serogroup C (Day 28 post-vaccination 2) | 47
  Serogroup Y (Day 28 post-vaccination 1) | 43
  Serogroup Y (Day 28 post-vaccination 2) | 48
  Serogroup W-135 (Day 28 post-vaccination 1) | 52
  Serogroup W-135 (Day 28 post-vaccination 2) | 55

3. Other Pre Specified Outcome: Number of Participants Reporting Solicited Injection-Site and Systemic Reactions Following Vaccination
Description: Solicited injection (Inj.) site reactions: Pain (Grade 1: no interference with activity, Grade 2: some interference, Grade 3: significant interference), erythema and swelling (Grade 1: >=25 to <=50 mm; Grade 2: >=51 to <=100 mm; Grade 3: >100 mm); Solicited systemic reactions: Fever (Grade 1: >=37.5 degree Celsius to <=38.4 degree Celsius, Grade 2: >=38.5 degree Celsius to <=38.9 degree Celsius, Grade 3: >=39.0 degree Celsius), headache, malaise and myalgia (Grade 1: no interference with activity, Grade 2: some interference, Grade 3: significant interference). Number of participants with any of the Grade 1, 2 or 3 solicited injection-site and systemic reactions and Grade 3 solicited injection-site and systemic reactions were reported.
Time Frame: Within 7 days post-vaccination 1, Within 7 days post-vaccination 2
Population: Safety analysis set included all participants who received at least 1 dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Menactra® Vaccine
Number analyzed (Participants) | 60
Participants
  Any Inj. site pain (post-vaccination 1) | 18
  Grade 3 Inj site pain (post-vaccination 1) | 0
  Any Inj site pain (post-vaccination 2): number analyzed (Participants) | 58
  Any Inj site pain (post-vaccination 2) | 17
  Grade 3 Inj site pain (post-vaccination 2): number analyzed (Participants) | 58
  Grade 3 Inj site pain (post-vaccination 2) | 0
  Any Erythema (post-vaccination 1) | 0
  Grade 3 Erythema (post-vaccination 1) | 0
  Any Erythema (post-vaccination 2): number analyzed (Participants) | 58
  Any Erythema (post-vaccination 2) | 0
  Grade 3 Erythema (post-vaccination 2): number analyzed (Participants) | 58
  Grade 3 Erythema (post-vaccination 2) | 0
  Any Swelling (post-vaccination 1) | 0
  Grade 3 Swelling (post-vaccination 1) | 0
  Any Swelling (post-vaccination 2): number analyzed (Participants) | 58
  Any Swelling (post-vaccination 2) | 0
  Grade 3 Swelling (post-vaccination 2): number analyzed (Participants) | 58
  Grade 3 Swelling (post-vaccination 2) | 0
  Any Fever (post-vaccination 1) | 1
  Grade 3 Fever (post-vaccination 1) | 0
  Any Fever (post-vaccination 2): number analyzed (Participants) | 58
  Any Fever (post-vaccination 2) | 1
  Grade 3 Fever (post-vaccination 2): number analyzed (Participants) | 58
  Grade 3 Fever (post-vaccination 2) | 0
  Any Headache (post-vaccination 1) | 5
  Grade 3 Headache (post-vaccination 1) | 0
  Any Headache (post-vaccination 2): number analyzed (Participants) | 58
  Any Headache (post-vaccination 2) | 5
  Grade 3 Headache (post-vaccination 2): number analyzed (Participants) | 58
  Grade 3 Headache (post-vaccination 2) | 0
  Any Malaise (post-vaccination 1) | 9
  Grade 3 Malaise (post-vaccination 1) | 0
  Any Malaise (post-vaccination 2): number analyzed (Participants) | 58
  Any Malaise (post-vaccination 2) | 3
  Grade 3 Malaise (post-vaccination 2): number analyzed (Participants) | 58
  Grade 3 Malaise (post-vaccination 2) | 0
  Any Myalgia (post-vaccination 1) | 12
  Grade 3 Myalgia (post-vaccination 1) | 0
  Any Myalgia (post-vaccination 2): number analyzed (Participants) | 58
  Any Myalgia (post-vaccination 2) | 11
  Grade 3 Myalgia (post-vaccination 2): number analyzed (Participants) | 58
  Grade 3 Myalgia (post-vaccination 2) | 0

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected from Day 0 (post-vaccination) up to 98 days at the longest.
Description: A solicited reaction is an AE that is prelisted in the electronic Case Report Form (eCRF) and considered to be related to vaccination. A solicited reaction is therefore an adverse drug reaction (ADR) observed and reported under the conditions (nature and time to onset) prelisted (i.e., solicited) in the eCRF.
  An unsolicited AE is an observed AE that does not fulfill the conditions prelisted in the eCRF in terms of symptom and/or time to onset post-vaccination.
Arm/Group | Menactra® Vaccine
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 32/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Menactra® Vaccine (N=60)
Headache (Nervous system disorders) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 18
Injection site pain (General disorders) | 25
Malaise (General disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.